CLINICAL TRIAL: NCT01618279
Title: Evaluation of Tryptase as a Biomarker of Coronary Heart Disease
Brief Title: Tryptase and Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 193_05/2012
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Acute Coronary Syndrome With ST Elevation on Electrocardiogram; Acute Coronary Syndrome Without ST Elevation on Electrocardiogram; Noncritical Coronary Artery Disease Coronary Stenosis Less Than 50 Per Cent; Aortic Aneurysms
Keywords: tryptase; coronary; stemi; nstemi
MeSH Terms: conditions — Aortic Aneurysm; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tryptase: Patients with clinical manifestations have been discovered and documented symptoms of coronary heart

SUMMARY:
The main aim of this study will evaluate differences in serum levels of tryptase in study population. Will be selected a number of 350 patients hospitalized for coronary heart disease.

DETAILED DESCRIPTION:
A series of scientific studies have evaluated the tryptase as a biomarker of coronary plaque instability, in the course of ischemic heart disease. Among these, the most recent and 'outcome' is better defined by Meixiang Xiang study, which has been conducted in 2011 on 270 patients. This study evaluated and compared the levels of tryptase in four populations:

1. acute myocardial infarction (31 subjects)
2. unstable angina (108 subjects)
3. stable angina (36 subjects)
4. coronary artery disease with coronary stenosis <50% (95 subjects). In this Chinese population the final evaluations have led to define the tryptase as a marker independent of instability of the atheromatous plaque.

In reference to the fact that there is still some correlation between tryptase and coronary plaque instability and clinical symptoms, we propose a verification study of the role of tryptase as a biomarker in acute coronary conditions by studying a large population of Italian subjects in the acute phase of pathology and follow up.

The work will be conducted on 4 patient population:

1. acute coronary syndrome with ST elevation on electrocardiogram;
2. acute coronary syndrome without ST elevation on electrocardiogram (acute myocardial infarction with ST-segment depression on electrocardiogram and unstable angina)
3. noncritical coronary artery disease with coronary stenosis <50%;
4. aortic aneurysms. Secondary endpoints will evaluate the role of tryptase in the event of major cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects aged 18 to 80 years
* patients with clinical manifestations have been discovered and documented symptoms of coronary heart disease
* all patients with these characteristics will necessarily have to sign the informed consent for inclusion in the study

Exclusion Criteria:

* patients with allergy symptoms in place (hives, uncontrolled asthma) autoimmune diseases, mastocytosis, hypereosinophilia, myelodysplastic syndrome, cancer, kidney failure
* those who deny consent to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Italian subjects in the acute phase of disease and follow up. The work will be on 4 patient populations:
  1. sindrome coronary acute ST elevation on electrocardiogram
  2. sindrome ACS without ST elevation on electrocardiogram (acute myocardial infarction with ST-segment depression on electrocardiogram and unstable angina)
  3. malattia critical coronary artery stenosis <50%
  4. aneurismi aorta.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
serum level of tryptase as a biomarker in coronary | 6 months
  dose level of serum tryptase already performed by venipuncture from diagnostic practices

SECONDARY OUTCOMES:
Tryptase and major cardiovascular events | 6 months
  correlation between the level of tryptase and probable major cardiovascular events (death, myocardial infarction or reinfarction and stroke)
Tryptase and major cardiovascular events | 6 months
  cut-off level of tryptase distinguishing between the study population and identified individuals at risk of major cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Elide Anna Pastorello, MD, Professor, Principal Investigator — Azienda Ospedaliera Ospedale Niguarda Ca' Granda
Locations (1):
- AO Osepdale Niguarda Ca' Granda, Milan, Italy

REFERENCES:
- [Background] Morici N, Farioli L, Losappio LM, Colombo G, Nichelatti M, Preziosi D, Micarelli G, Oliva F, Giannattasio C, Klugmann S, Pastorello EA. Mast cells and acute coronary syndromes: relationship between serum tryptase, clinical outcome and severity of coronary artery disease. Open Heart. 2016 Sep 27;3(2):e000472. doi: 10.1136/openhrt-2016-000472. eCollection 2016. PMID 27752333
- [Background] Pastorello EA, Morici N, Farioli L, Di Biase M, Losappio LM, Nichelatti M, Lupica L, Schroeder JW, Stafylaraki C, Klugmann S. Serum tryptase: a new biomarker in patients with acute coronary syndrome? Int Arch Allergy Immunol. 2014;164(2):97-105. doi: 10.1159/000360164. Epub 2014 Jun 14. PMID 24943670
- [Background] Pastorello EA, Farioli L, Losappio LM, Morici N, Di Biase M, Nichelatti M, Schroeder JW, Balossi L, Klugmann S. Serum tryptase detected during acute coronary syndrome is significantly related to the development of major adverse cardiovascular events after 2 years. Clin Mol Allergy. 2015 Jun 2;13(1):14. doi: 10.1186/s12948-015-0013-0. eCollection 2015. PMID 26038676
- [Background] Losappio LM, Mirone C, Chevallard M, Farioli L, De Luca F, Pastorello EA. Tryptase as a marker of severity of aortic valve stenosis. Clin Mol Allergy. 2018 Aug 7;16:17. doi: 10.1186/s12948-018-0095-6. eCollection 2018. PMID 30093839